CLINICAL TRIAL: NCT01408251
Title: Agreement Between Arterial, Central Venous, and Peripheral Venous Lactate in the Intensive Care Unit
Brief Title: Agreement Between Arterial, Central Venous, and Peripheral Venous Lactate Measurements in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Richard Treger/Principal Investigator, VA Greater Los Angeles Healthcare System
Other Study IDs: 193070
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Acid-base Analysis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to see if blood obtained from a vein (smaller blood vessel) can be used instead of blood obtained from an artery (larger blood vessel).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU and requiring both an arterial line and central venous line as prt of their clinical care

Exclusion Criteria:

* Patient did not desire to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Unit patients requiring both an arterial line and central venous line as part of their clinical care
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Treger, M.D., Principal Investigator — VA Greater Los Angeles Healthcare System